CLINICAL TRIAL: NCT01007578
Title: An Open-Labeled Multicenter Study to Investigate Plasma Levels and Catheter Tolerability Following Application of Paclitaxel Coated Balloon Catheter in Patients With Stenotic, or Occluded Femoro-Popliteal Arteries Due to Atherosclerosis
Brief Title: Drug-Eluting Balloon Catheters and the Treatment of Peripheral Arterial Occlusive Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-4601-900
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Peripheral Arterial Disease; Stenotic Femoro-popliteal Arteries; Occluded Femoro-popliteal Arteries; Atherosclerosis
Keywords: Paclitaxel; Paclitaxel-coated balloon catheters; Peripheral arterial occlusive disease (PAOD); Plasma levels; Femoral artery; Popliteal artery; Peripheral arterial disease (PAD) including stenotic or occluded femoro-popliteal arteries due to atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel treatment (Experimental): Paclitaxel-coated balloon catheter angioplasty treated subjects
  Interventions: Device: Paclitaxel-coated balloon catheter angioplasty

INTERVENTIONS:
Device: Paclitaxel-coated balloon catheter angioplasty — Paclitaxel-coated balloon catheters for the treatment of peripheral arterial occlusive disease (POAD) of the femoro-popliteal arteries

SUMMARY:
The purpose of this study is to determine plasma levels of paclitaxel and catheter tolerability subsequent to treating patients with peripheral arterial occlusive disease (PAOD) with paclitaxel-coated balloon catheters.

DETAILED DESCRIPTION:
This is an open-labeled multicenter study to investigate plasma levels and catheter tolerability following application of paclitaxel-coated balloon catheter angioplasty in patients with stenotic or occluded femoro-popliteal arteries due to atherosclerosis. Safety will be assessed by changes in blood cell (leukocytes, neutrophils and thrombocytes) counts, and changes in serum biochemistry parameters. Tolerability will be assessed by adverse event occurences related to the paclitaxel-coating and/or device by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met all of the following criteria for inclusion in the study:

  1. Clinically stable patients with PAOD disease, Rutherford stage 1, 2, 3, 4, or 5.
  2. Occlusion up to 5 cm or a ≥70% diameter stenosis of up to 32 cm length in the Arteria (A.) femoralis superficialis or A. popliteal, documented by angiography prior to intervention.
  3. Age: >18 years.
  4. Guide wire may successfully advance across the lesion.
  5. Patient was eligible for an operative vascular intervention in case of complications.
  6. Informed consent was signed by patient after information of possible alternatives.
  7. Women of childbearing potential must had negative results in serum pregnancy test and use a reliable method of contraception.

     Exclusion Criteria:
* Patients who met any of the following exclusion criteria were not included in the study:

  1. Previous treatment at the same location.
  2. Close affiliation with the investigational site; e.g., a close relative of the Investigator, dependent person (e.g., employee or student of the investigational site).
  3. Acutely occurring symptoms (within the last 6 weeks) with a lysis or an operation as a therapeutic option.
  4. Potential loss of leg due to ischemia.
  5. Distal blood flow over less than one lower leg blood vessel.
  6. Aneurysm of intended treatment blood vessel.
  7. Women of child bearing potential (and up to 2 years postmenopausal) without a negative pregnancy test.
  8. Manifest hyperthyreosis or latent hyperthyreosis without previous blocking (sodium phosphonate).
  9. Blood platelet count <100.000/mm^3 or >700.000/mm^3, leukocyte count <3.000/mm^3.
  10. Known intolerance or contra-indication to aspirin, heparin, clopidogrel, abciximab, paclitaxel, or stainless steel, and known intolerance to contrast agents which cannot be adequately pre-treated.
  11. Illnesses (cancer, liver diseases, myocardial insufficiency) leading to protocol deviations and a reduced life expectancy (<2 years).
  12. Renal insufficiency with serum creatinine over 2.0 mg/dL.
  13. Diabetes mellitus with additional metformin therapy.
  14. Significant gastrointestinal hemorrhage in the previous 6 months.
  15. History of hemorrhagic diathesis or coagulopathy or rejection of blood transfusions due to religious or other reasons.
  16. Patient who received any investigational device or combination product for the intended indication within the 30 days prior to entering this study.
  17. Patient who had previously participated in another study using a paclitaxel coated catheter.
  18. Non-compliant or incapable patients to participate in the study (patients unable to speak or understand German language), patients not willing to answer questions regarding the study via telephone, patients rejecting an electronic storage of their patient information, or imprisoned patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-09-15 (Actual); Primary Completion 2007-12-15 (Actual); Study Completion 2007-12-15 (Actual)

PRIMARY OUTCOMES:
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty at baseline | Baseline
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty 0.5 hours post-procedure | 0.5 hours post-procedure
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty 1 hour post-procedure | 1 hour post-procedure
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty 2 hours post-procedure | 2 hours post-procedure
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty 4 hours post-procedure | 4 hours post-procedure
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty 8 hours post-procedure | 8 hours post-procedure
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty 1 week post-procedure | 1 week post-procedure
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty 2 weeks post-procedure | 2 weeks post-procedure
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty 3 weeks post-procedure | 3 weeks post-procedure
Plasma levels of paclitaxel in patients with stenotic or occluded femoro-popliteal arteries following application of paclitaxel-coated balloon catheter angioplasty 4 weeks post-procedure | 4 weeks post-procedure

SECONDARY OUTCOMES:
Changes in blood cell counts as measure of safety at baseline | Baseline
Changes in blood cell counts as measure of safety 0.5, 1, 2, 4, 8 and 24 hours post-procedure | 0.5, 1, 2, 4, 8 and 24 hours post-procedure
Changes in blood cell counts as measure of safety 1, 2, 3, and 4 weeks post-procedure | 1, 2, 3, and 4 weeks post-procedure
Changes in serum biochemistry parameters as measure of safety at baseline | Baseline
Changes in serum biochemistry parameters as measure of safety 0.5, 1, 2, 4, 8 and 24 hours post-procedure | 0.5, 1, 2, 4, 8 and 24 hours post-procedure
Changes in serum biochemistry parameters as measure of safety 1, 2, 3, and 4 weeks post-procedure | 1, 2, 3, and 4 weeks post-procedure
Number of participants with adverse events (AEs) as a measure of safety | From randomization until end of study, up to 4 months
Number of participants with serious adverse events (SAEs) as a measure of safety | From randomization until end of study, up to 4 months
Number of participants with adverse device effects (ADEs) as a measure of safety | From randomization until end of study, up to 4 months
Number of participants with adverse events (AEs) judged as possible/probable/definitely related to the paclitaxel coating and/or device by the investigator as a measure of tolerability | From randomization until end of study, up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Herz-Zentrum Bad Krozingen, Bad Krozingen, Germany